CLINICAL TRIAL: NCT04474106
Title: The Effect of Extracorporeal Shock Wave Therapy (ESWT) in Acute Traumatic Complete (AIS A) and Incomplete (AIS B-D) Cross-sectional Lesions on Motor and Sensory Function Within Six Months After Injury: A Two-arm Three-stage Adaptive, Prospective, Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: NEUROwave - Extracorporeal Shock Wave Therapy (ESWT) in Acute Traumatic Complete (AIS A) and Incomplete (AIS B-D) Cross-sectional Lesions on Motor and Sensory Function Within Six Months After Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AUVA (Other)
Responsible Party: Principal Investigator, Wolfgang Schaden, Deputy Medical Director of Austrian Workers´ Compensation Board (AUVA), AUVA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEUROwave
Record Dates: First submitted 2020-06-30; First posted 2020-07-16 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Acute Traumatic Spinal Cord Injury

STUDY DESIGN:
Intervention Model Description: Two-arm three-stage adaptive, prospective, multi-center, randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stratified block randomization with a block size of four and a 1:1 allocation will be used to assign participants to one of two groups (treatment vs. placebo). Three neurological levels of injury will be used for stratification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT (Experimental): The extracorporeal shockwave therapy is applied once at the level of lesion and 5 segments above and below; or below the occiput (in lesions higher than C6) and above the sacrum (in lesions lower than T12). In addition, the ESWT is applied to the soles of both feet on the medial side of the plantar surface. The ESWT is applied as soon as possible within 48 hours post-injury.
  Interventions: Device: Shock waves
- Control (Sham Comparator): In the control group, the same procedure is performed, but without the device emitting extracorporeal shock waves using a dummy head.
  Interventions: Device: dummy head

INTERVENTIONS:
Device: Shock waves — The shockwave generator orthogold 100® generates high-energy acoustic waves that behave much like other sound waves except that they have much greater pressure and energy. As with sound waves, Spark Waves® can easily travel great distance as long as the acoustic impedance stays the same.
  Arms: ESWT
Device: dummy head — The shockwave generator orthogold 100® will be used in combination with a dummy head, to Refrain shock waves
  Arms: Control

SUMMARY:
It has been hypothesized that there are two mechanisms of acute traumatic spinal cord injury (SCI): the primary mechanical damage and the secondary injury due to additional pathological processes initiated by the primary injury. Neurological damage due to laceration, contusion, distraction or compression of the spinal cord is called ''primary injury''. This mechanical injury leads to a cascade of biochemical and pathological changes, described as ''secondary injury'', which occurs minutes to weeks after the initial trauma and causes further neurological deterioration. This secondary cascade involves vascular changes, an inflammatory response, neurotoxicity, apoptosis and glial scarring, and further compromises neurological impairment after traumatic spinal cord injury. Edema, ischemia and loss of autoregulation continue to spread bi-directionally from the initial lesion along the spinal cord for up to 72 hours after the trauma.

It has been postulated that the damage caused by the primary injury mechanism is irreversible and therapeutic approaches in recent years have focused on modulating the secondary injury cascade.

Researchers found significantly greater numbers of myelinated fibers in peripheral nerves after a single ESWT application in an experimental model on rats after a homotopic nerve autograft into the sciatic nerve.

In another study a spinal cord ischemia model in mice was performed. ESWT was applied immediately after surgery and the treated animals showed a significantly better motor function and decreased neuronal degeneration compared to the control group within the first 7 days after surgery.

Researchers investigated the effect of low-energy ESWT for the duration of three weeks on a thoracic spinal cord contusion injury model in rats. Animals in the ESWT group demonstrated significantly better locomotor improvement and reduced neuronal loss compared to the control animals at 7, 35, and 42 days after contusion.

It has been postulated previously, that ESWT improves the metabolic activity of various cell types and induces an improved rate of axonal regeneration.

ESWT might be a promising therapeutic strategy in the treatment of traumatic SCI.

The underlying study aims to investigate the effect of ESWT after acute traumatic spinal cord injury in humans within 48 hours of trauma in order to intervene in the secondary injury phase with the objective to reduce the extent of neuronal damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute traumatic spinal injuries who are awake, responsive, and oriented at admission
* Patients from the age of 18 years
* Admission to hospital within 24 hours after injury
* Written consent to participate in the study
* Participation in the Austrian Spinal Cord Injury Study (ASCIS)-Registry (only for the Austrian hospitals)

Exclusion Criteria:

* Patients who cannot cooperate or are not capable to give consent to participate
* Serious traumatic brain injuries that prevent accurate participation in study procedures and/or adequacy of informed consent Participation in other interventional clinical trials
* Serious concomitant injuries that prevent the neurological initial assessment
* Preexisting neurological conditions that affect the primary endpoint of the study and potentially mask or reduce the therapeutic effect of the ESWT application
* High dose administration of corticosteroids
* Complete spinal cord transection
* Patients with pacemakers or implantable defibrillators
* Patients who are using devices which are sensitive to electromagnetic radiation
* (potential) Pregnancy
* Patients with tumors
* Patients with severe coagulation disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in total motor scores (TMSC) = TMSC after 6 month minus TMSC at baseline | day 0 to 6 month
  greater improvement in motor and sensory function (the AIS grade) can be achieved in patients after spinal trauma (AIS A-D) by applying a single extracorporeal shockwave therapy compared to the control group.

SECONDARY OUTCOMES:
American Spinal Injury Association (ASIA) Impaiment Scale (AIS) grade | day 0 to 6 month
  the AIS grade ranges from AIS A to AIS D, whereby AIS A are complete lesions and AIS B-D represent incomplete lesions
degree of spasticity | day 0 to 6 month
  self-rated degree of spasticity according to Penn Spasm Frequency Scale (PSFS); the scale ranges from 0 to 4, whereby 0 refers to no spasticity and 4 refers to more than 10 spasms per hour
Walking ability (yes/no) | day 0 to 6 month
  walking ability is being assessed using different walking tests as part of standard clinical routine: Walking Index for Spinal Cord Injury (WISCI) II, Timed up and go test (TUG), 10 Meter-Timed-Walk, 6 Minute-Walk-Test
Urological function | day 0 to 6 month
  Urological function will be assessed by several questions which should be answered with yes or no:
  * Permanent catheter: yes/no
  * Sensation of urinary bladder filling: yes/no
  * Documentation of the first attempt of bladder emptying: pos/neg, date
  * Self-catheterization: yes/no
  * Do you feel sensory innervation of the external genitalia (penis / labia)?
  * Do you feel the change of the catheter or manipulations on the catheter?
  * Do you feel the urge to defecate?
  * Do you feel stool evacuation?
  * Male patients: Have you had an erection since your injury?
  * Female patients: Have you felt sexually aroused since your injury?
Plantar reflex (left/right: yes/no) | day 0 to 6 month
  The plantar reflex (also called Babinski Test) will be performed separately on each foot to assess if pathological reflexes are present.
Independence in everyday life | day 0 to 6 month
  of patients is assessed with the Spinal Cord Independence Measure (SCIM II)
adverse events (AEs) | day 0 to 21 days
  The number of study related adverse events (AEs) are measured according to NCI CTCAE, version 5.0.
Nine-Hole Peg Test (NHPT) (if feasible) | day 0 to 6 month
  An evaluation of hand motor function is assessed in those patients who have their lesions above the level T5
Grasp and Release Test (GRT) | day 0 to 6 month
  An evaluation of hand motor function is assessed in those patients who have their lesions above the level T5
Pinch grip: yes/no | day 0 to 6 month
  An evaluation of hand motor function is assessed in those patients who have their lesions above the level T5
Clenched grip: yes/no | day 0 to 6 month
  An evaluation of hand motor function is assessed in those patients who have their lesions above the level T5
Pencil grip: yes/no | day 0 to 6 month
  An evaluation of hand motor function is assessed in those patients who have their lesions above the level T5
Lumbrical grip: yes/no | day 0 to 6 month
  An evaluation of hand motor function is assessed in those patients who have their lesions above the level T5

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Schaden, Dr., Principal Investigator — AUVA
Locations (15):
- Austria (15):
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Rehazentrum Bad Häring, Bad Häring
  - Landeskarnkenhaus Feldkirch, Feldkirch
  - Unfallkrankenhaus Graz, Graz
  - Rehazentrum Tobelbad, Graz
  - Unfallkrankenhaus Klagenfurt, Klagenfurt
  - Rehazentrum Weißer Hof, Klosterneuburg
  - Unfallkrankenhaus Linz, Linz
  - Unfallkrankenhaus Salzburg, Salzburg
  - Universitätsklinik für Orthopädie und Traumatologie, Salzburg
  - Unfallkrankenhaus St. Pölten, Sankt Pölten
  - Universitätsklinik Wien, AKH, Vienna
  - Unfallkrankenhaus Meidling, Vienna
  - Unfallkrankenhaus Lorenz Böhler, Vienna
  - SMZ Ost, Donauspital Abteilung für Unfallchirurgie, Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leister I, Mittermayr R, Mattiassich G, Aigner L, Haider T, Machegger L, Kindermann H, Grazer-Horacek A, Holfeld J, Schaden W. The effect of extracorporeal shock wave therapy in acute traumatic spinal cord injury on motor and sensory function within 6 months post-injury: a study protocol for a two-arm three-stage adaptive, prospective, multi-center, randomized, blinded, placebo-controlled clinical trial. Trials. 2022 Apr 1;23(1):245. doi: 10.1186/s13063-022-06161-8. PMID 35365190